CLINICAL TRIAL: NCT00259038
Title: A Phase II, Dose Escalation Evaluation of the Pharmacokinetic and Hemodynamic Effects of Carperitide in Subjects With Congestive Heart Failure
Brief Title: Evaluation of the Effects of Carperitide in Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-0-162
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Heart Failure, Congestive; Heart Decompensation; Left Ventricular Failure; Myocardiopathies; Systolic or Diastolic Left Ventricular Dysfunction
Keywords: Carperitide; Atrial Natriuretic Peptide; Treatment efficacy; Safety; Heart failure, Congestive; Pulmonary Artery Catheterization
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Systolic Murmurs; Ventricular Dysfunction, Left | interventions — NPPA protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Experimental Drug (Experimental)
  Interventions: Drug: Carperitide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carperitide
  Other Names: human recombinant atrial natriuretic peptide
  Arms: Experimental Drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the safety and efficacy of intravenous infusion of carperitide using pressure measurements inside the heart and great vessels and measuring carperitide concentration in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Is hospitalized with congestive heart failure (CHF)
* Has a Swan-Ganz catheter inserted for CHF management and has pulmonary capillary wedge pressure 18 mmHg or higher

Exclusion Criteria:

* Has had a heart transplant
* Requires mechanical ventilation or mechanical circulatory support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2004-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pulmonary capillary wedge pressure (PCWP) | at 3 hours following initiation of study drug infusion

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Pavlovic-Surjancev, MD, PhD, Study Director — Astellas Pharma US, Inc.
Locations (32):
- United States (28):
  - Huntsville, Alabama
  - Los Angeles, California
  - Orange, California
  - San Diego, California
  - Bay Pines, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Springfield, Illinois
  - Covington, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Albany, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Amarillo, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Tacoma, Washington
  - Madison, Wisconsin
- Canada (4):
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
  - Saint Foy, Quebec